CLINICAL TRIAL: NCT03560102
Title: Efficacy of Magnetic Resonance-guided High Intensity Focused Ultrasound for the Ablation of Breast Cancer: Correlation Between MRI and Histology. Single-Center, Single-Arm, Non-Randomized Trial
Brief Title: Efficacy of Magnetic Resonance-guided High Intensity Focused Ultrasound for the Ablation of Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01282 (BASEC); 2017-MD-0021 (Other: Swissmedic)
Record Dates: First submitted 2018-05-14; First posted 2018-06-18 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer, Invasive Ductal
MeSH Terms: conditions — Carcinoma, Ductal, Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-HIFU treatment (Experimental): Patients with breast cancer and scheduled surgical resection (lumpectomy or mastectomy) will be treated with Philips Sonalleve® MR-HIFU Breast Therapy System prior to surgery in a treat& resect model
  Interventions: Device: Philips Sonalleve® MR-HIFU Breast Therapy System

INTERVENTIONS:
Device: Philips Sonalleve® MR-HIFU Breast Therapy System — The breast tumor lesion of qualified study patients will be treated with MR-HIFU under procedural sedation with Propofol and Ketamine.

SUMMARY:
The purpose of the study is to evaluate the efficacy of a dedicated Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU) unit in ablating breast cancer by comparing MR imaging and pathologic specimen after resection.

Single-center, single-arm, non-randomized trial

DETAILED DESCRIPTION:
The dedicated MR-HIFU unit has been shown to be safe and feasible to ablate breast tissue.

The planned study should address the possibility to completely ablate breast cancer with the dedicated breast MR-HIFU unit. The result of the MR-HIFU therapy should be monitored by imaging (contrast enhanced MRI) as well as with histopathological correlation after surgery.

The patient population would consist of female patients with proven breast cancer scheduled for surgical lumpectomy or mastectomy.

The idea is to evaluate a minimal invasive method to treat breast cancer as a potential alternative to surgical resection in the future

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* World Health Organization (WHO) performance status≤ 2
* Body weight ≤ 80 kg
* Biopsy proven invasive breast cancer with a size of ≤3.0cm (TNM classification: cT1-2 N0-2 MX ).
* Histological type of tumor: invasive ductal carcinoma (IDC)
* Patient is scheduled for surgical resection of tumor at study site
* Tumor location within the reach of the HIFU transducers with the patient in prone position; distance from skin and pectoral muscle to the tumor ≥ 1.0 cm.
* Target breast fits in the cup of the dedicated MR-HIFU breast system

Exclusion Criteria:

* neoadjuvant systemic therapy
* prior radiotherapy in target breast
* contraindications for MRI
* contraindication for application of gadolinium-based contrast agent
* contraindication for procedural sedation analgesia
* macro-calcifications in or around the targeted tumor
* scar tissue or surgical clips in the direct path of the ultrasound beams
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug/device within the 30 days preceding and during the present study,
* Previous enrolment into the current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Binkert, MD, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enroled: 06JAN2020 Last patient completed: 05FEB2020
Pre-assignment Details: Due to difficulties in recruitment only 2 patients were screened for inclusion and only 1 patient met inclusion criteria and was enrolled in the study.
Period: Overall Study
Arm/Group | MR-HIFU Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MR-HIFU Treatment
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 1
Height [Mean (Standard Deviation); unit: cm] | 163 (0)
Weight [Mean (Standard Deviation); unit: kg] | 65 (0)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of MRI as Method for Assessment of Quantitative Treatment Success (Correlation With Results of the Histopathological Analysis Performed as Reference Method)
Description: Quantitative assessment: Correlation between MRI and histopathology results (volume of necrosis)
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: percentage of histopathological result
Arm/Group | MR-HIFU Treatment
Number analyzed (Participants) | 1
percentage of histopathological result | 168 (0)

2. Secondary Outcome: Assessment of Treatment Efficacy
Description: Effective treatment is defined as complete necrosis (100%) of targeted tumor including safety margin (>1mm) (histopathological analysis).
  Safety margin: measurement of smallest margin on histology and measurement of smallest margin on MRI. Parameter: Percentage of necrosis including safety margin
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: percentage of necrosis of targeted tumor
Arm/Group | MR-HIFU Treatment
Number analyzed (Participants) | 1
percentage of necrosis of targeted tumor | 3.9 (0)

3. Other Pre Specified Outcome: Incidence of Adverse Events [Safety and Tolerability of the Treatment]
Description: Adverse events, general:
  Patients will be asked to report information about adverse events at each time point of the study. Information about time of onset, duration, resolution, action to be taken assessment of intensity, relationship with study treatment will be collected.
  Assessment of additional predefined safety parameters:
  - Skin changes, assessment in physical examination: presence/absence of redness, burn
  * Palpation breast: lump (mobility of lump related to skin: yes/no)
  * Pain, reported by patient
Time Frame: Day 0, 3, 8
Measure: Count of Participants; unit: Participants
Arm/Group | MR-HIFU Treatment
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Follow-up: Day 2, Day 8 (End of study)
Arm/Group | MR-HIFU Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT03560102/Prot_SAP_000.pdf